CLINICAL TRIAL: NCT01841567
Title: A Multi-centre, Post CE-mark, Open Investigation to Evaluate the Performance of a Flexible Self-adherent Absorbent Dressing Coated With a Soft Silicone Layer After Hip or Knee Arthroplasty
Brief Title: Post Market Clinical Follow-up Study
Acronym: MxB Po01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxB Po01
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2013-12

CONDITIONS: Hip or Knee Surgery
Keywords: hip; knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dressing (Other)
  Interventions: Device: Mepilex border post. op; Device: Mepilex border post op

INTERVENTIONS:
Device: Mepilex border post. op
Device: Mepilex border post op

SUMMARY:
The overall rationale for this study is to evaluate the clinical performance potential for Mepilex Border Post-Op in the ability to minimise the risk of blistering, maceration and less dressing change due to high absorption capacity. This study is a part of Post Market Clinical Follow-Up (PMCF).

ELIGIBILITY:
Inclusion Criteria

1. Age 45 years
2. Have an expected total length of stay of 4 or more days
3. Undergoing elective primary arthroplasty of the hip or knee
4. Undergoing hip surgery with a standard access
5. Give their written informed consent to participate

Exclusion Criteria

1. Dressing size does not fit the incision area
2. Known allergy hypersensitivity to any of the components of the dressing
3. Multi-trauma
4. Undergoing arthroplasty due to tumour
5. Fractures
6. Wound at the surgical site prior to surgery
7. Neurological deficit of operated side
8. Subject has documented skin disease at time of enrolment, as judged by the investigator
9. Previously enrolled in the present investigation
10. Subject included in other ongoing investigation at present, as judged by the investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Zarghooni, Dr. Med, Principal Investigator — University Hospital Koln
Locations (1):
- universitätsklinikum Köln, Cologne, Köln, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Dressing: Mepilex border post. op
  Mepilex border post op
Period: Overall Study
Arm/Group | Dressing
Started | 60
Completed | 57
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dressing
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 22
Region of Enrollment [Number; unit: participants]
  Germany | 60

OUTCOME MEASURES:

1. Primary Outcome: Minimize the Risk of the Development of Blistering.
Description: Number of participants without blisters at study visit
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Dressing
Number analyzed (Participants) | 60
participants | 60

2. Secondary Outcome: Number of Participants Rated 'Very Good to Excellent' for Comfort, Conformability and the Acceptability of the Dressing.
Description: The comfort, conformability and the acceptability of the dressing were measured on all visit in the study, by a study nurses. The patient had to answer questions regarding, the size of the dressing, shape of the dressing, Visibility beneath the dressing, ease of the application of the dressing, ease of removal of the dressing, overall experience of the use of the dressing, notice any pain at dressing change, Comfort of their dressing, overall experience of their dressing. The patient could chose between 1 Good, 2 Very good, 3 Excellent.In most cases, the patient chose very good to excellent for both hip and knee surgery
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Dressing
Number analyzed (Participants) | 60
participants | 60

3. Secondary Outcome: Comfort, Comformability, Acceptability of the Dressing
Time Frame: 7 days

4. Secondary Outcome: Pain Evaluation
Time Frame: 7 days

5. Secondary Outcome: Overall Cost Regarding Dressing Wear Time
Time Frame: 7 days

ADVERSE EVENTS:
Arm/Group | Dressing
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dressing (N=60)
•Cardiac disorders (Cardiac disorders) | 1 (1) — suspicion of heart attack, no relation to the study product
surgical and medical procedures (Surgical and medical procedures) | 1 (1) — reoperation due to implantdislocation, no relation to the study product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other